CLINICAL TRIAL: NCT04467307
Title: Comparison of Symptoms and Findings and Short-term Results After Bronchoscopy in Patients With and Without the Foreign Body in Children Under 5 Years Old Who Underwent Bronchoscopy With Suspicion of Foreign Body Aspiration. A Prospective Study.
Brief Title: Comparison of Patients With and Without Foreign Body Aspiration After Bronchoscopy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Ahmet Gökhan Güler, Department of pediatric surgery, Kahramanmaras Sutcu Imam University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2020/02-02
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Foreign Body Aspiration, Blood Gas, Bronchoscopy
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foreign body aspiration. (Active Comparator): Patients undergoing bronchoscopy with suspicion of foreign body aspiration. There is a foreign body in the bronchoscopy performed on these patients and it is the treated group.
  Interventions: Device: Rigit bronchoscopy
- Group with no foreign body aspiration (Active Comparator): Patients undergoing bronchoscopy with suspicion of foreign body aspiration, but there is no foreign body in bronchoscopy.
  Interventions: Device: Rigit bronchoscopy

INTERVENTIONS:
Device: Rigit bronchoscopy — After general anesthesia, the airway is checked with a rigid bronchoscope suitable for the age. If there is a foreign body, it is removed by forceps.

SUMMARY:
To compare patients under 5 years of age with foreign body aspiration and without foreign body aspiration with radiological and blood gas results.

DETAILED DESCRIPTION:
Foreign body aspiration in children is a serious cause of mortality and morbidity. It is a preventable and treatable disease. Difficulties in diagnosis arise in non-radiopaque foreign body aspirations. Recently, when there is a suspicious history, bronchoscopy is recommended. Bronchoscopy is used to both diagnose and treat foreign body aspiration. Bronchoscopy seems to continue to be performed in suspicious cases until a method to establish a definitive diagnosis of foreign body aspirations before the operation is invented. In our study, to compare patients under 5 years of age with foreign body aspiration and without foreign body aspiration with radiological and blood gas results.

ELIGIBILITY:
Inclusion Criteria:

Suspected foreign body aspiration

Exclusion Criteria:

infection, trauma

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Foreign body aspiration | 1 week
  The presence of a foreign body in the airway by bronchoscopy, radiological findings, blood gas

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, Onikisubat, Turkey (Türkiye)